CLINICAL TRIAL: NCT00985543
Title: Pharmacokinetics of Plasma Lopinavir/Ritonavir Over a 12 Hour Dosing Interval Following Administration of 400/100, 200/150, and 200/50 mg Twice Daily to HIV-negative Healthy Volunteers
Brief Title: Pharmacokinetics of Lopinavir/Ritonavir at Three Different Doses.
Acronym: ENCORE3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Marta Boffito, Chelsea and Westminster Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHECR-ENCORE3
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: HIV; ART; HAART; Pharmacokinetics; Lopinavir/ritonavir; Lower dose selection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LPV/r 400/100 mg (Active Comparator): Lopinavir/ritonavir 400/100 mg twice daily (2 heat-stable 200/50 mg tablets twice daily (BID))
  Interventions: Drug: lopinavir/ritonavir
- LPV/r 200/150 mg (Experimental): Lopinavir/ritonavir 200/150 mg twice daily (1 heat-stable 200/50 mg tablet BID plus 1 ritonavir 100 mg capsule BID)
  Interventions: Drug: lopinavir/ritonavir
- LPV/r 200/50 mg (Experimental): Lopinavir/ritonavir 200/50 mg twice daily (1 heat-stable 200/50 mg tablet BID)
  Interventions: Drug: lopinavir/ritonavir

INTERVENTIONS:
Drug: lopinavir/ritonavir — Each participant received three sequential doses of lopinavir/ritonavir: 400/100 mg twice daily (2 heat-stable 200/50 mg tablets BID), 200/150 mg twice daily (1 heat-stable 200/50 mg tablet BID plus 1 ritonavir 100 mg capsule BID), and 200/50 mg twice daily (1 heat-stable 200/50 mg tablet BID). Each dosing phase lasted for 7 days and each phase was separated by a 7-day wash-out period.
  Other Names: Meltrex; Ritonavir

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of plasma lopinavir/ritonavir over a 12-hour dosing interval, following administration to male and female HIV-negative healthy volunteers of:

1. Lopinavir/ritonavir 400/100 mg twice daily
2. Lopinavir/ritonavir 200/150 mg twice daily
3. Lopinavir/ritonavir 200/50 mg twice daily

DETAILED DESCRIPTION:
Data during the development of lopinavir/ritonavir showed that lower drug doses had similar efficacy to the standard dose of 400/100mg twice daily. Lower drug doses are also associated with limited toxicity and cost.

The purpose of this study is to assess the pharmacokinetics of plasma lopinavir/ritonavir following administration to male and female HIV-negative volunteers of 400/100mg, 200/150mg and 200/50mg lopinavir/ritonavir twice daily. Each dosing phase will last for 7 days and each phase will be separated by a 7-day wash-out period. Pharmacokinetic evaluations will be made over a 12-hour interval at the end of each dosing phase.

Healthy subjects as determined by their medical history and physical examinations will be eligible to participate in the study. HIV-positive subjects will not be recruited as there is a risk that HIV-resistant mutations will be selected by an experimentally reduced dose of lopinavir/ritonavir. There is no reason to presume that there is any meaningful difference in the metabolic processing of lopinavir/ritonavir between HIV-infected and HIV-uninfected people.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria within 28 days prior to the baseline visit:

  1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
  2. Male or non-pregnant, non-lactating females
  3. Between 18 to 65 years, inclusive
  4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
  5. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month after the study

Exclusion Criteria:

1. Any significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B core and/or C antibodies and/or hepatitis B surface antigen
4. Positive blood screen for HIV-1 and/or 2 antibodies
5. Current or recent (within 3 months) gastrointestinal disease
6. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
7. Exposure to any investigational drug or placebo within 3 months of first dose of study drug
8. Consumption of grapefruit, or Seville oranges or any grapefruit or Seville orange containing product within one week of first dose of study drug and for the duration of the study
9. Use of any other drugs, including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
10. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 30 days after the end of the treatment period
11. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MD PhD, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- St Stephen's Centre, Chelsea and Westminster Hospital, London, United Kingdom

REFERENCES:
- [Derived] Jackson A, Hill A, Puls R, Else L, Amin J, Back D, Lin E, Khoo S, Emery S, Morley R, Gazzard B, Boffito M. Pharmacokinetics of plasma lopinavir/ritonavir following the administration of 400/100 mg, 200/150 mg and 200/50 mg twice daily in HIV-negative volunteers. J Antimicrob Chemother. 2011 Mar;66(3):635-40. doi: 10.1093/jac/dkq468. Epub 2010 Dec 17. PMID 21172791

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All participants were given three sequential doses of lopinavir/ritonavir: lopinavir/ritonavir 400/100mg twice daily (2 heat-stable 200/50mg tablets BID), lopinavir/ritonavir 200/150mg twice daily (1 heat-stable 200/50mg tablet BID plus 1 ritonavir 100mg capsule BID), lopinavir/ritonavir 200/50mg twice daily (1 heat-stable 200/50mg tablet BID). Each dosing phase lasted for 7 days and each phase was separated by a 7-day wash-out period. Pharmacokinetic evaluations were made over a 12-hour interval at the end of each dosing phase.
Period: Overall Study
Arm/Group | All Study Participants
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22

OUTCOME MEASURES:

1. Primary Outcome: Plasma Lopinavir/Ritonavir Concentrations as Measured by the Area Under the Curve (AUC 0-12h).
Description: Pharmacokinetics of plasma lopinavir/ritonavir over a 12-hour dosing interval following administration of lopinavir/ritonavir 400/100mg, 200/150mg and 200/50mg twice daily.
Time Frame: at the end of each 7-day dosing phase
Population: 22 participants completed the three sequential dosing phases and pharmacokinetic evaluations as per protocol. The same 22 participants are in the analysis population for each lopinavir/ritonavir dose (arm).
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | LPV/r 400/100 mg | LPV/r 200/150 mg | LPV/r 200/50 mg
Number analyzed (Participants) | 22 | 22 | 22
ng.h/mL | 99599 [87180 to 113787] | 73603 [65121 to 83191] | 45146 [39251 to 51927]
Statistical Analysis 1: Comparison: LPV/r 400/100 mg vs LPV/r 200/150 mg vs LPV/r 200/50 mg; Dosing regimens lopinavir/ritonavir 200/150mg BID (Phase 2) and lopinavir/ritonavir 200/50mg BID (Phase 3) will be considered equivalent to lopinavir/ritonavir 400/100mg BID (Phase 1) if the 90% confidence interval (CI) for the mean AUC0-12h ratio and maximum concentration (Cmax) ratio lie between 0.80 and 1.25; Test type: Non-Inferiority or Equivalence — Results are considered statistically significant at p<0.05 or when 90% confidence intervals do not cross the value 1. No adjustments are made for multiple comparisons; p < 0.05, maximum likelihood regression

2. Secondary Outcome: Adverse Events
Description: Number of reported adverse events, severity of adverse events and relationship to study drug was assessed by questions, physical examination and laboratory parameters. Adverse event data was used to assess the safety and tolerability of low lopinavir/ritonavir doses.
Time Frame: Up to 11 weeks from screening to final study visit
Population: as for outcome 1
Measure: Number; unit: number of adverse events
Arm/Group | LPV/r 400/100 mg | LPV/r 200/150 mg | LPV/r 200/50 mg
Number analyzed (Participants) | 22 | 22 | 22
number of adverse events | 27 | 2 | 4

ADVERSE EVENTS:
Time Frame: Up to 11 weeks from screening visit until the participant's final study visit.
Description: Any adverse event that occurred after the reporting period that the PI assesses as possibly, probably or definitely related to the study drug was also reported.
Groups:
- All Study Participants: All participants were given three sequential doses of lopinavir/ritonavir: lopinavir/ritonavir 400/100mg twice daily (2 heat-stable 200/50mg tablets BID), lopinavir/ritonavir 200/150mg twice daily (1 heat-stable 200/50mg tablet BID plus 1 ritonavir 100mg capsule BID), lopinavir/ritonavir 200/50mg twice daily (1 heat-stable 200/50mg tablet BID). Each dosing phase lasted for 7 days and each phase was separated by a 7-day wash-out period.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 15/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=22)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 4 (4)
Headache (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not publish or otherwise disseminate the conclusions of the Study, including all or any part of the Results without the prior written consent of the Sponsor, such consent not to be unreasonably withheld or delayed. Any publication or other dissemination of the conclusions of the Study by the PI shall not occur until the Sponsor has published the conclusions of the Study.